CLINICAL TRIAL: NCT05876325
Title: Leveraging Medical Legal Partnerships to Enhance Patient-Centered, Team-Based Cost Conversations With Pediatric Oncology Patients and Families
Brief Title: Financial and Insurance Assistance- Oncology Financial and Legal Navigation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean Edward (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor-Investigator, Jean Edward, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 57238
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Financial Stress; Pediatric Cancer
Keywords: Financial toxicity; Hardship; Cost conversations; FINassist
MeSH Terms: conditions — Financial Stress; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Financial Navigation and Insurance Assistance (FINassist) (Experimental): FINassist is a comprehensive oncology financial and legal navigation program in oncology care
  Interventions: Other: FINassist Patient; Other: FINassist Caregiver

INTERVENTIONS:
Other: FINassist Patient — The FINassist intervention provides access to social, financial and legal services over the duration of 12 months or until issues are resolved
Other: FINassist Caregiver — The FINassist intervention provides access to social, financial and legal services over the duration of 12 months or until issues are resolved

SUMMARY:
The overall objective of this study was to develop and evaluate FINassist (Financial and Insurance Navigation Assistance), a patient-centered, interdisciplinary team-based oncology financial and legal navigation program. The program leverages Medical Legal Partnerships to enhance cost of care conversations with pediatric oncology patients and caregivers. FINassist optimizes the team-based care model by integrating clinicians, social workers, financial navigators, and legal advocates who work in tandem to enhance cost of care conversations with patients and caregivers, identify and intervene on patient socio-legal needs, and advocate for system-level changes.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of patients who have any cancer or hematologic disorder diagnosis at the DanceBlue Pediatric Hematology/oncology clinic at Kentucky Children's hospital
* Patients with childhood cancers and/or hematologic disorders at the DanceBlue Pediatric Hematology/oncology clinic at Kentucky Children's hospital
* 18 years and older

Exclusion Criteria:

* Unable to provide consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants enrolled | 12 months
  Feasibility was defined as 60% or higher enrolled participant retention and resolution of financial or legal issue (based on existing oncology financial navigation studies)
FINassist Adherence | through issue resolution up to 12 months
  Adherence is defined by the percentage of participants that maintain communication with the team and provide documents necessary for issue resolution
FINassist Retention | through study completion up to 12 months
  percentage of participants that complete both pre and post-intervention surveys
FINassist Acceptability assessed by 5-item survey | Post intervention at 12 months
  Acceptability is measured using a 5 item post-intervention survey of relevance, helpfulness, convenience, recommendation to others, and value. Ratings on a scale from 0 to 10 where a higher score means greater acceptability
Change in Total Financial Toxicity | Baseline and post intervention, approximately 12 weeks
  Measured using the COmprehensive Score for financial Toxicity (COST) tool, a measure that describes the financial distress experienced by cancer patients. Scores range from 0-44 with a higher score representing better financial well-being.
Change in Participant Quality of Life (physical and mental) | Baseline and post intervention, approximately 12 weeks
  Measured using the 10-item PROMIS® (Patient-Reported Outcomes Measurement Information System) Parent Proxy Global Health scale. A 7-item summary assessment of a child's self-reported health with higher scores representing better quality of life. Values range from 7-35, with higher scores representing better health.
Change in Participant Quality of Life (Depression) | Baseline and post intervention, approximately 12 weeks
  Measured using the 6-item Patient-Reported Outcomes Measurement Information System PROMIS® Depression Short Form. Scores range from 6 to 30. Higher scores indicate more of the construct being measured.
Change in Participant Quality of Life (Anxiety) | Baseline and post intervention, approximately 12 weeks
  Measured using the 4-item Patient-Reported Outcomes Measurement Information System PROMIS® Anxiety short form. Scores range from 4 to 20. Higher scores indicate more of the construct being measured.
Change in Patient-Provider Trust | Baseline and post intervention, approximately 12 weeks
  Measured using the the Health Care Relationship (HCR) Trust Scale. The HCR-Trust scale is scored from 0 to 4 with a maximum score of 52. Higher scores represent more trust in healthcare providers
Resolution of Socio-legal Issue | 12 months
  Number of participants that resolved a legal or financial case as a result of FINassist
Change in PROMIS Parent Proxy Global Health | Baseline and post intervention, approximately 12 weeks
  used to measure child QOL (when applicable), with summary scores for proxy measures of global health, pain interference, and fatigue Overall evaluation of physical, mental health, and social health.
Change in PROMIS Parent Proxy Pain Interference | Baseline and post intervention, approximately 12 weeks
  used to measure child QOL (when applicable), with summary scores for proxy measures of global health, pain interference, and fatigue Consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities.
Change in PROMIS Parent Proxy Fatigue | Baseline and post intervention, approximately 12 weeks
  used to measure child QOL (when applicable), with summary scores for proxy measures of global health, pain interference, and fatigue Range of symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion.

SECONDARY OUTCOMES:
Number of Participants Receiving Financial Benefit | 12 months
  financial benefit defined as economic hardship avoided or decreased public/government income

CONTACTS AND LOCATIONS:
Overall Officials: Jean Edward, PhD, RN, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky DanceBlue Pediatric Hematology/oncology clinic, Lexington, Kentucky, United States

REFERENCES:
- [Derived] Edward J, Northrip KD, Rayens MK, Welker A, O'Farrell R, Knuf J, Fariduddin H, Costich J, D'Orazio J. Financial-legal navigation reduces financial toxicity of pediatric, adolescent, and young adult cancers. JNCI Cancer Spectr. 2024 Apr 30;8(3):pkae025. doi: 10.1093/jncics/pkae025. PMID 38552323